CLINICAL TRIAL: NCT04302506
Title: The Correlative Cohort Study on the Clinical Features and Prognosis of Drug-induced Liver Injury
Brief Title: Correlative Cohort Study on the Clinical Features and Prognosis of Drug-induced Liver Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Director of Hepatology Division 2, Beijing Ditan Hospital
Other Study IDs: DTXY025
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Drug-induced Liver Injury
Keywords: Drug-induced liver injury; Chronic; regression analysis; ROC curve; Joint diagnosis
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with drug-induced liver injury: Patients who underwent liver biopsy and were diagnosed with drug-induced liver injury were diagnosed as DILI.

SUMMARY:
This was a retrospective study of a clinical observational cohort. The patients were admitted and definitely diagnosed by liver biopsy as drug-induced liver injury from September 2014 to September 2019, in the Second Department of Liver Disease, Beijing Ditan Hospital Affiliated to Capital Medical University were enrolled, and these patients also met the RUCAM score and were clinically diagnosed as DILI. Baseline clinical data and follow-up biochemical data at 3, 6, and 12 months were collected. SPSS software was used to analyze the characteristics of clinical data and the dynamic changes of biochemical indicators. Logistic regression was used to analyze the risk factors associated with the chronicity of DILI. Bivariate Logistic regression model and ROC curve were used to obtain the clinical indicators for combined diagnosis of chronicity of DILI patients. To investigate the clinical features and prognostic factors of drug-induced liver injury.

DETAILED DESCRIPTION:
This was a retrospective study of a clinical observational cohort. The patients were admitted and definitely diagnosed by liver biopsy as drug-induced liver injury from September 2014 to September 2019, in the Second Department of Liver Disease, Beijing Ditan Hospital Affiliated to Capital Medical University were enrolled, and these patients also met the RUCAM score and were clinically diagnosed as DILI. Baseline clinical data and follow-up biochemical data at 3, 6, and 12 months were collected. SPSS software was used to analyze the characteristics of clinical data and the dynamic changes of biochemical indicators. Logistic regression was used to analyze the risk factors associated with the chronicity of DILI. Bivariate Logistic regression model and ROC curve were used to obtain the clinical indicators for combined diagnosis of chronicity of DILI patients. To investigate the clinical features and prognostic factors of drug-induced liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Have a clear history of taking drugs (Chinese herbal medicine and dietary supplements, NSAIDs, cardio-cerebrovascular drugs, anti-interference drugs, anti-tuberculosis drugs, hormone drugs and others);
* All patients were examined by liver biopsy Patients with clear diagnosis of drug-induced liver injury and clinical diagnosis of DILI who meet the RUCAM score.

Exclusion Criteria:

* Combined with various liver diseases, such as viral hepatitis (hepatitis A, B, C, D, E), alcoholic hepatitis, autoimmune hepatitis, metabolic hepatitis, non-alcoholic fatty liver disease;
* Combining other viral infections that may lose liver function, such as Epstein-Barr Virus (EBV), Cytomegalovirus (CMV), and Human Immunodeficiency Virus (HIV);
* Mental illness;
* Evidence of liver tumors (liver cancer or alpha-fetoprotein> 100 ng / ml).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Department of Hepatology Division 2, Beijing Ditan Hospital, Capital Medical University was admitted and a liver biopsy was performed from 2014.9 to 2019.9. The patients were clearly diagnosed with drug-induced liver injury. These patients also met the RUCAM score and were diagnosed as DILI.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
The rate of chronicity | 48 weeks
  Chronic rate of drug-induced liver injury

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatology Division 2, Beijing Ditan Hospital, Beijing, Beijing Municipality, China